CLINICAL TRIAL: NCT03740646
Title: Primary-Pneumocystis Infection: Pneumocystis Jirovecii Detection in Nasopharyngeal Aspirates From Symptomatic Infants
Brief Title: Pneumocystis Primary Infection in Non-immunosuppressed Infants
Acronym: CAPRI-PC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CAPRI-PC( 29BRC18.0052)
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Diseases; Fever
Keywords: Bronchiolitis; Nasopharyngeal aspirates
MeSH Terms: conditions — Lung Diseases; Fever; Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal aspirates with or without Pneumocystis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the prevalence of P. jirovecii in nasopharyngeal aspirations of neonates and infants hospitalized for symptomatic respiratory infection.

DETAILED DESCRIPTION:
It is recognized that primary infection with Pneumocystis, an opportunistic and transmissible fungus, occurs early in childhood. Early investigations of primary infection considering the detection of P. jirovecii in respiratory specimens suggests that primary infection in infants without immunodeficiency could be either asymptomatic or symptomatic. The infection may be identified as an apparently benign respiratory infection evolving on its own, but may also be contemporaneous with another viral or bacterial respiratory infection. In addition, there are little data available on the genotypic characteristics of P. jirovecii in infants developing primary infection.

In this context, the project will focus on the detection of P. jirovecii in hospitalized infants, presented with symptoms, and without overt immunodeficiency. The prospective collection of biological, clinical and epidemiological data in these infants will make it possible to identify risk factors for the acquisition of the fungus and to address its role in symptoms and clinical presentation. A second focus will be on the identification and comparison of genotypes in infants developing primary infection and in immunocompromised adults developing PPC or colonized by the fungus. These two approaches are the necessary steps to address the putative role of these patient populations (infants and adults) in the human reservoir of the fungus. A third focus will be the detection and genotypic identification of P. jirovecii in infants and the exhaled air of infants in their environment. The potential role of infants as potential infectious sources may be determined.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic newborns and infants who underwent NPAs for microbiological diagnoses

Exclusion Criteria:

* asymptomatic newborns and infants, newborns and infants who did not undergo NPAs, infants > 12 months or children > 2 years; newborns and infants whose parents did not accept to participate

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: symptomatic newborns and infants who underwent NPAs for microbiological diagnoses
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Pneumocystis presence or not in nasopharyngeal specimens from newborns and infants | At patient inclusion
  The main biological parameter which will be measured will be the positive or negative result of P. jirovecii detection in nasopharyngeal apsirate specimens from non-immunosuppressed newborns and infants. The prevalence of P. jirovecii comtemporary with first contacts with the fungus will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: NEVEZ Gilles, MD PhD, Principal Investigator — Brest University Hospital, Brest, France
Locations (1):
- CHRU de Brest, Brest, France